CLINICAL TRIAL: NCT05680051
Title: A Prospective, Multi-center, Randomized, Parallel Controlled Clinical Trial of Drug Coated Balloon Under the Guidance of OCT in the Treatment of Acute ST-segment Elevation Myocardial Infarction
Brief Title: DCB Under the Guidance of OCT in STEMI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Institute of Cardiovascular Epidemiology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HenanICE202208
Record Dates: First submitted 2022-12-14; First posted 2023-01-11 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Acute ST-segment Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Drug-Eluting Stents

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Drug-coated Balloon (Lepu Medical Technology (Beijing) Co.,Ltd.)
  Interventions: Device: Drug-eluting balloon
- Control group (Active Comparator): Drug Eluting Stent(Microport Medical)
  Interventions: Device: Drug-eluting stent

INTERVENTIONS:
Device: Drug-eluting balloon — Drug eluting balloon was used in the experimental group
  Arms: Experimental group
Device: Drug-eluting stent — Drug eluting stent was used in the control group
  Arms: Control group

SUMMARY:
Acute ST segment elevation myocardial infarction (STEMI) has a high disability mortality rate, and timely reperfusion treatment can significantly reduce the mortality of patients. Emergency PCI is the preferred strategy for STEMI treatment recommended by domestic and international guidelines. The long-term existence of stents can never completely avoid the formation of thrombosis in the stents and affect the relaxation and contraction of criminal blood vessels. Drug coated balloon provides a new concept and technology of interventional therapy for coronary artery disease in the form of "intervention without implantation". Through balloon dilation of local blood vessels to release anti proliferative drugs to coronary artery wall and inhibit intimal hyperplasia, it can not only treat serious coronary artery disease, improve coronary blood supply and vascular function, but also not leave permanent implants in the blood vessels; The main pathogenesis of STEMI is thrombosis based on the rupture or erosion of coronary atheromatous plaque. In terms of pathophysiological mechanism, drug coated balloons are also suitable for STEMI patients without obvious thrombosis or severe dissection after full pretreatment. The two-dimensional lumen images obtained by traditional coronary angiography can not directly reflect the vessel wall, so we can not evaluate the actual size of the vessel, plaque characteristics and the effect of intervention through coronary angiography; Optical coherence tomography (OCT) uses near-infrared scanning to produce high-resolution tissue microscopic images with a resolution of up to 10 μ m. It can clearly observe the three-layer structure of coronary artery, find abnormal intima structure, and more clearly identify thrombosis, dissection, plaque erosion or collapse in coronary artery, providing more valuable information for optimizing interventional treatment. Therefore, the application of drug coated balloon under the guidance of OCT in STEMI can provide a more accurate and optimized diagnosis and treatment scheme for STEMI patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75
2. Definitely diagnosed as acute ST segment elevation myocardial infarction according to diagnostic criteria
3. Time of onset ≤ 12h
4. Voluntary signing of informed consent
5. After pretreatment, the culprit vessel participates in stenosis ≤ 30%, no type C (or OCT shows that the dissection involves the middle membrane, and the angle is ≥ 90 degrees) or above, no hematoma, and no obvious thrombus (TIMI thrombus load rating ≤ 2)

Exclusion Criteria:

1. Time of onset>12h
2. Those who are allergic to contrast agents, aspirin tablets and Tigrilol tablets;
3. Active bleeding or recent bleeding history
4. Cardiogenic shock and long-term cardiopulmonary resuscitation;
5. The life span is expected to be less than 12 months
6. Angiography showed left main trunk lesion;
7. Angiography shows patients with in stent restenosis
8. Patients who the investigator thinks may affect the normal progress of the study or cannot cooperate well with the study or may cause obvious risks, such as alcoholics or drug abusers, cancer, serious liver, kidney, lung, endocrine (such as uncontrolled diabetes or thyroid disease), nervous or blood system diseases;
9. Known or suspected pregnancy (baseline ß - hCG pregnancy test must be conducted for women in childbearing period), women in menstrual period.
10. The criminal blood vessel has C-type or above dissection after pretreatment, and there is coronary hematoma.
11. After pretreatment, criminal vessels still have obvious thrombus residues (TIMI thrombus load grade ≥ 3)
12. OCT confirms that the criminal lesion is caused by plaque erosion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Late lumen loss rate | 10 months after discharge.

SECONDARY OUTCOMES:
Revascularization rate of target lesions | 10 months after discharge.
Target vessel revascularization rate | 1 month after discharge, 3 months after discharge, 6 months after discharge, 10 months after discharge.
Major Adverse Cardiovascular Events | 1 month after discharge, 3 months after discharge, 6 months after discharge, 10 months after discharge.
Cardiovascular death | 1 month after discharge, 3 months after discharge, 6 months after discharge, 10 months after discharge.
Recurrent acute myocardial infarction | 1 month after discharge, 3 months after discharge, 6 months after discharge, 10 months after discharge.
  Time-to-onset for recurrent acute myocardial infarction, as ascertained according to follow-up
Stroke | 1 month after discharge, 3 months after discharge, 6 months after discharge, 10 months after discharge.
  Time-to-onset for stroke, as ascertained according to follow-up
All cause of death | 1 month after discharge, 3 months after discharge, 6 months after discharge, 10 months after discharge.
Unstable angina | 1 month after discharge, 3 months after discharge, 6 months after discharge, 10 months after discharge.
  Time-to-onset for unstable angina, as ascertained according to follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Central China Cardiovascular Hospital, Zhengzhou, Henan, China